CLINICAL TRIAL: NCT03763084
Title: Impact of Oral Acetaminophen Analgesia on Postoperative Delirium and Long-term Survival in Elderly Patients After Non-cardiac Surgery: A Randomized Controlled Trial
Brief Title: Impact of Acetaminophen on Postoperative Delirium Elderly Patients After Non-cardiac Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018071027
Record Dates: First submitted 2018-12-02; First posted 2018-12-04 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-11

CONDITIONS: Acetaminophen; Delirium in Old Age
Keywords: acetaminophen; analgesia; delirium
MeSH Terms: conditions — Agnosia; Delirium | interventions — Acetaminophen; Sufentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- acetaminophen (Experimental): For patients randomized to OVA group, OVA 500mg was given every 8 hours for the first 48 hours postoperatively. Numeric Pain Rating Scale pain score is assessed every 15 minutes during the 1 hour of ICU stay and when needed.
  Interventions: Drug: Acetaminophen
- Sufentanil (Active Comparator): Sufentanil injection 500μg /10ml in normal saline, total volume 50 ml.Constant infusion dosage is 0.05μg/kg/h. Numeric Pain Rating Scale pain score is assessed every 15 minutes during the 1 hour of ICU stay and when needed.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Acetaminophen — For patients in the acetaminophen group, oral acetaminophen supplemented dexmedetomidine sedation will be provided after surgery.
  Arms: acetaminophen
Drug: Sufentanil — For patients in the control group, sufentanil supplemented dexmedetomidine sedation will be provided after surgery.
  Arms: Sufentanil

SUMMARY:
To investigate the impact of acetaminophen analgesia on the frequency of postoperative delirium and 28 days mortality in elderly patients after noncardiac surgery.

DETAILED DESCRIPTION:
Background: Delirium is a common complication following surgery contributes to adverse outcomes, including increased mortality and morbidity, longer length of ICU stays, prolonged mechanical ventilation, and costlier hospitalizations. Previous studies showed that, the incidence of delirium for seniors patients admitted to ICU can reach up to 58%-75.6% depending on the patient population and screening instrument. The current protocols for perioperative opioid use and postoperative pain management may influence the occurrence of delirium. We hypothesize that the use of oral acetaminophen (OVA) may lead to reduced opioid consumption and decreased incidence of postoperative delirium.

Objectives: To investigate the impact of acetaminophen analgesia on the frequency of postoperative delirium and 28 days mortality in elderly patients after noncardiac surgery.

Study design: A randomized and controlled trial. Setting: Departments of critical care medicine of tertiary hospital (Xiangya) in China.

Patients: 164 elderly patients (≥ 65 years) who are scheduled to admitted to ICU after major surgery (predicted duration ≥ 2 hours) Intervention: For patients in the acetaminophen group, oral acetaminophen supplemented dexmedetomidine sedation will be provided after surgery. For patients in the control group, sufentanil supplemented dexmedetomidine sedation will be provided after surgery. the other analgesia drugs will be provided as back up in study group.

Primary outcome: Early primary endpoint is the frequency of delirium in the first 5-days post-surgery. Secondary endpoints include biomark and NeuroMonitoring of delirium, 28days and in-hospital mortality, length of stay days in ICU and hospital, complication in hospital.

Predicted duration of the study: 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to ICU after non-cardiac surgery for any reasons；
2. Report having moderate to severe acute pain as determined by a pain score ≥ 5 from the 11-point Numeric Pain Rating Scale (NPRS) scale after postsurgery；
3. Able to take oral medication or by stomach tube；
4. Provide written informed consent.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded.

  1. Preoperative history of schizophrenia, epilepsy, Parkinsonism, or myasthenia gravis;
  2. Inability to communicate in the preoperative period because of coma, profound dementia or language barrier;
  3. Brain injury or neurosurgery;
  4. Severe hepatic dysfunction (eg, aspartate aminotransferase, alanine aminotransferase, or bilirubin greater than or equal to 3.0 times the upper limit of normal), active hepatic disease, evidence of clinically significant liver disease, or other condition (eg, alcoholism, cirrhosis, or hepatitis) that suggests the potential for an increased susceptibility to hepatic toxicity with study drug exposure.
  5. Subject has a positive test result for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methamphetamine, methadone, or methylenedioxy-methamphetamine) at Screening.
  6. Subject has participated in another clinical study within 30 days prior to day-of-surgery or plans to participate in another clinical study while concurrently enrolled in this study.
  7. Subject has a history of any drug allergy, hypersensitivity, or intolerance to acetaminophen or morphine or to any of the excipients in the IV or oral formulations used.
  8. Subject has intra- or postoperative complications, which in the view of the investigator, makes the subject unsuitable for the participation of the study.
  9. Subject has a history of any drug allergy, hypersensitivity, or intolerance to acetaminophen or opioid or to any of the excipients in the IV or oral formulations used.
  10. Unable to take medications orally or by stomach tube

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of delirium | within the first 5 postoperative days
  evaluate the occurence of delirium by using Confusion Assessment Method for The Intensive Care Unit (CAM-ICU)

SECONDARY OUTCOMES:
Effectiveness of analgesia | during postoperative days 1-5
  to assess the effect of analgesia by using Numerical Rating Scale (NRS)；This method is composed of 0 to 10, a total of 11 Numbers. Patients with 0 to 10 this digital describe pain intensity, the greater the number the pain degree is more serious.0 painless, 1 ~ 3 mild pain (pain does not affect sleep), 4 ~ 6 moderate pain, 7 ~ 9 severe pain (couldn't sleep), 10 severe pain. We should ask the patient pain degree, tag, or let the patient draw one of the most can represent their own pain degree of digital.
Length of days in ICU and hospital stay after surgery | from day 1 after surgery to discharge (up to 24 weeks)
  evaluate the length of days in ICU and hospital stay from postoperative to discharge
Incidence of non-delirium complications | with 28 days after surgery
  Incidence of non-delirium complications with 28 days after surgery
All-cause28-day mortality | day 28 after surgery
  All-cause28-day mortality
life-Quality evaluation of 28-day survivors | day 28 after surgery
  evaluate the quality of life by using the world health organization quality of life measurement scale(WHOQOL-BREF). WHOQOL-BREF contains 26 items, summarizes the physiological, psychological, social relations, the environment in the field of four content.Consists of two independent analysis problem items: question 1 (G1) ask individual about their quality of life of the general subjective feeling, question 2 (G4) individual asked the total subjective feeling bout their own health. Domain scores are the positive (i.e., the higher the score, the better the quality of life).Field scoring through the calculation of average of their entries 4 times. and patients will be assessed via phone call if they are discharged before day 28 after surgery
Cognitive function of 28-day survivors | day 28 after surgery
  evaluate the cognitive function of 28-day survivors by using modified version of the telephone questionnaire for cognitive function questionnaire (TICS-m);It contains 21 items, total score 50 points, can be divided into three parts: the memory part (score 20), directional force (score 13), the capablity of language, and pay attention (score 17). TICS -m total score 50 points, scored < 28 divided into dementia, 28 and 33 were divided into mild cognitive dysfunction, ≥33 were divided into normal. Patients will be assessed via phone call if they are discharged before day 28 after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China